CLINICAL TRIAL: NCT05561621
Title: Prediction of Non-motor Symptoms in Fully Ambulatory MS Patients Using Vocal Biomarkers
Acronym: COMMITMENT
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Audeering GMBH (Industry); Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: DLF5177
Record Dates: First submitted 2022-09-27; First posted 2022-09-30 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Digital Biomarker; Non-Motor symptoms; Fatigue; Cognition; Depression; Voice Analysis
MeSH Terms: conditions — Multiple Sclerosis; Fatigue; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with relapsing MS
  Interventions: Other: Voice analysis
- Healthy controls
  Interventions: Other: Voice analysis

INTERVENTIONS:
Other: Voice analysis — Voice analysis

SUMMARY:
The investigator will set up a study evaluating vocal biomarkers in people with MS in order to identify persons with non-motor symptoms: depression, cognitive deterioration, and fatigue. Up to now, to the best of the investigator's knowledge, there is no study reporting the use of vocal biomarkers to predict these three non-motor symptoms in people with MS.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing MS
* Age over 18
* EDSS < 4.0
* Capability of written informed consent

Exclusion Criteria:

* Not fluent in german language
* Relapse or Steroids per os/intra venous < 4 weeks prior to examination
* KM enhancing lesion in MRI < 4 weeks prior to examination
* Other previous disease affecting the speech
* Pregnant patients
* Mental disability and not able to understand the protocol and study tasks in german languagePatients with greater physical and cognitive disability or history of major depressive disorder and suicide attempt/suicidal thoughts
* Patients with sleep disorders and comorbidities associated with extreme fatigue (e.g., fibromyalgia)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with relapsing MS and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Identification of a voice signature that separates between pwMS with and without fatigue | One year

SECONDARY OUTCOMES:
Identification of a voice signature that separates between pwMS with and without cognitive impairment | One year
Identification of a voice signature that separates between pwMS with and without depression | One year

CONTACTS AND LOCATIONS:
Overall Officials: Helly Hammer, Principal Investigator — Inselspital, University Hospital Bern
Locations (1):
- Inselspital University Hospital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No